CLINICAL TRIAL: NCT02293694
Title: A 12-month Open-label Randomized Controlled Trial to Evaluate Sayana® Press Suitability for at Home Subcutaneous Self-injection Procedures in Adult Women
Brief Title: Sayana® Press Self-injection Study in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 631917-1
Record Dates: First submitted 2014-11-10; First posted 2014-11-18 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Contraception
Keywords: DMPA-SC: depo medroxyprogesterone acetate sub-cutaneous; DMPA-IM: depo medroxyprogesterone acetate intramuscular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-injection (Active Comparator): Women randomized to this arm will be trained to self-inject Sayana Press at home every three months
  Interventions: Drug: Sayana Press
- provider injection (Active Comparator): Women randomized to this arm will received Sayana press from a family planning provider every three months.
  Interventions: Drug: Sayana Press

INTERVENTIONS:
Drug: Sayana Press — Sayana® Press is a subcutaneous formulation of depot medroxyprogesterone acetate (DMPA) in a prefilled, auto-disabled injection system called Uniject
  Other Names: depot medroxyprogesterone acetate (DMPA)

SUMMARY:
The feasibility of Sayana Press self-injection and the potential for this practice to increase contraceptive continuation has never been assessed in family planning programs in low-resource settings. The Malawi Ministry of Health (MOH) and the United States Agency for International Development (USAID) Malawi Mission requested the Advancing Partners and Communities (APC) project to assess self-injection of Sayana Press to inform their decision-making for procurement of Sayana Press and distribution through the health system in Malawi.

DETAILED DESCRIPTION:
Sayana® Press is a subcutaneous formulation of depot medroxyprogesterone acetate (DMPA) in a prefilled, auto-disabled injection system called Uniject (Pfizer, Inc., USA). Sayana Press was registered with the Medicines and Health Care Products Regulatory Agency (MHRA) and several other national regulatory agencies. The addition of this method is anticipated to aid in improving provision of family planning services in low-resource settings. As such, Sayana Press could be particularly useful in a country such as Malawi where injectable contraception is the most common method used. DMPA clients and providers are ready to explore the potential of self-injection of Sayana Press. A study conducted in a large family planning clinic in Edinburgh, Scotland found self-administration of DMPA-SC feasible and associated with similar continuation rates and satisfaction to clinician-administered DMPA-IM. A non-comparison study conducted in Planned Parenthood clinics in Florida found continuation of self-injected DMPA-SC high (74%) at the fourth injection. Participants in this study reported the injection to be easy and convenient and were likely to recommend self-administration to other women. Moreover, on September 29, 2014 Pfizer submitted a request to the MHRA to change the Sayana Press label to include self-injection.

If self-injection is found feasible, the results from this research will inform self-injection training materials, messages for providers and clients, and future scale-up efforts in Malawi and elsewhere in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

Age 18-40, inclusive

* In general good health (participant verbally reports she feels well)
* Able to understand and willing to sign an informed consent document
* Willing to give contact information for follow-up
* Agree to have follow-up visits/interviews
* Willing to be randomized to the self-injection arm or provider-administered injection arm
* Menstrual period started within the past 7 days (for new DMPA users)
* Meet eligibility criteria for receiving DMPA per WHO Medical Eligibility Criteria (MEC)

Exclusion Criteria:

Pregnancy

* Plans to become pregnant in the next 12 months
* Plans to relocate outside the study area in the next 12 months
* Any condition (social or medical) which in the opinion of the investigator would make study participation unsafe or would interfere with adherence to study requirements or complicate data interpretation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 735 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
To compare continuation rates between women who self-inject Sayana Press compared to women who receive Sayana Press injection from a provider | up to 12 months
  Discontinuation of Sayana Press measured at enrollment and every three months through one year

SECONDARY OUTCOMES:
To compare reported side effects between the two study groups | up to 12 months
  Women's reported side effects
To compare pregnancy rates between the two study groups | 12 months
  Frequencies of pregnancies in the two groups reported during the final

OTHER OUTCOMES:
To describe experiences of women who self-inject Sayana Press | 12 months
  Self-injectors' reported experiences (e.g., using, storing, and disposing of Sayana Press)
To describe experiences and recommendations of family planning providers who train women to self-inject Sayana Press | 12 months
  Providers' reported experiences and recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Holly Burke, Ph.D., Study Director — FHI 360
Locations (1):
- College of Medicine, Department of Community Health, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burke HM, Chen M, Packer C, Fuchs R, Ngwira B. Young Women's Experiences With Subcutaneous Depot Medroxyprogesterone Acetate: A Secondary Analysis of a One-Year Randomized Trial in Malawi. J Adolesc Health. 2020 Nov;67(5):700-707. doi: 10.1016/j.jadohealth.2020.03.038. Epub 2020 May 7. PMID 32389457
- [Derived] Burke HM, Chen M, Buluzi M, Fuchs R, Wevill S, Venkatasubramanian L, Dal Santo L, Ngwira B. Effect of self-administration versus provider-administered injection of subcutaneous depot medroxyprogesterone acetate on continuation rates in Malawi: a randomised controlled trial. Lancet Glob Health. 2018 May;6(5):e568-e578. doi: 10.1016/S2214-109X(18)30061-5. Epub 2018 Mar 8. PMID 29526707